Effect of intravenous administration of 20% Mannitol on the Optic Nerve Sheath Diameter (ONSD) in patients with raised intracranial



pressure.

Approval no: 360(6-11)E^2/075/76

Date: 24 Feb, 2019

# 1. Proposal Title:

Effect of intravenous administration of 20% Mannitol on the Optic Nerve Sheath Diameter (ONSD) in patients with raised intracranial pressure.

# 2. Project summary:

This is a prospective observational cross-sectional study which will determine the extent of change brought in the optic nerve sheath diameter by the intravenous administration of 20% Mannitol in patients with raised intracranial pressure. The studied patient will be those above the age of 18 years with traumatic brain injury, acute stroke or intracranial hemorrhage, with the features of elevated intracranial pressure as diagnosed by clinical findings, ONSD value > 5 mm and under 20% Mannitol osmotherapy, admitted in the intensive care unit of our institution. Written informed consent will be taken and after the eligibility criteria are met, epidemiological data including age, sex, weight, BMI at the time of admission will be recorded. Measured baseline observational values including optic nerve sheath diameter, mean arterial pressure will also be recorded. Observational variables will be measured after 30 minutes, 60 minutes and 120 minutes following the intravenous administration of 20% Mannitol. The data will be tabulated and analysis performed with SPSS software. The primary outcome will be the change in optic nerve sheath diameter, while the correlation between these variables will also be interpreted.

#### 3. Introduction

Raised intracranial pressure is a common incidence and complication in critically ill patients. There have been intense studies and research for understanding the underlying patho-physiology and treatment. Much of our understanding of the intracranial pressure is based on the Monro-Kellie hypothesis which states that the sum of intracranial volumes of blood, brain, CSF and other components is constant, and that an increase in any one of these must be offset by an equal decrease in another or else the pressure increases. The normal ICP is defined as 5 to 15 mmHg (7.5-20 cmH<sub>2</sub>O). Under normal conditions the brain is able to auto-regulate its blood flow. Cerebral perfusion pressure (CPP) defined by the equation CPP = MAP - ICP, is the single-most important determinant of this auto-regulation. Within a CPP ranging from 50-150 mmHg, the auto-regulation is intact. However during any insult/injury this ability of the brain may be impaired or absent thus leading to an unregulated change in ICP. Trauma, intracranial hemorrhage, intracranial tumors and ischemic stroke are the major causes of such insult and raised intracranial pressure.<sup>2</sup> Prompt diagnosis and treatment of elevated intracranial pressure is the cornerstone of management in TBI, intracranial hemorrhages and acute stroke and has been associated with poor outcomes. Care based on ICP monitoring has been proved to be associated with frequency of good recovery and favorable outcome.<sup>3</sup> Such monitoring can be invasive or non-invasive. Currently, invasive ICP monitoring is the gold standard. External ventricular drainage and micro-transducer ICP monitoring devices are the commonly used modes for ICP monitoring. However there are various hazards (infection and hemorrhage) of such invasive procedures and few studies have shown no such difference in outcomes with or without invasive monitoring.<sup>4,5</sup>

There have been various validated modes of non-invasive ICP monitoring. Trans-cranial Doppler ultrasonography (TCD), optic nerve sheath diameter (ONSD), tympanic membrane displacement and fundoscopic examinations have been proposed as being surrogates to invasive ICP monitoring.<sup>3,4</sup>, There have been many studies comparing the use of invasive against the use of non-invasive modes of ICP monitoring. Among these Optic nerve sheath diameter (ONSD) can be taken as the simplest mode with high positive and negative predictive values on detecting rise in intracranial pressure.<sup>6</sup> It's correlation with invasively measured intracranial pressure and imaging findings has also been validated<sup>7</sup> and used extensively in diagnosing episodes of raised intracranial pressure in emergency departments, intensive and neurosurgical units.<sup>8</sup>

The optic nerve is part of the central nervous system and therefore surrounded by the dural sheath. Between the sheath and the white matter is a small 0.1-0.2 mm subarachnoid space which communicates with the intracranial subarachnoid space. In cases with raised intracranial pressure the pressure is also transmitted into this sheath and expansion occurs. This expansion is appreciable via various imaging modalities like CT scans, MRI and ultrasonographic imaging. The feasibility and simplicity of this measurement by ultrasonography has made it a efficient tool in diagnosing and monitoring in acute care setup. The major drawbacks are the inter-observer variation in measurement and conditions that may confound the finding such as tumors, inflammation, grave's disease and sarcoidosis. Change in ONSD measurements performed before and after interventions including hyperventilation, drainage of CSF, administration of Mannitol, tracheal manipulation and lumbar puncture appear to correlate well with the induced change in ICP.<sup>6, 7</sup>

The incidence of elevated ICP is more than 50% in patients with ICP ranging as high as 80% in patients with traumatic brain injury. <sup>10, 11</sup> The fundamental goal of management in TBI is based on managing ICP, maintaining adequate CPP and is based upon the Monro-Kellie doctrine and cerebral autoregulation. <sup>11</sup> Similarly incidence of raised intracranial pressure in patient with intracranial hemorrhage ranges from 36% to 80%. <sup>12</sup> Malignant cerebral edema leading to raised intra-cranial pressure is a major cause of adverse outcome in patients with acute ischemic stroke with an incidence of 10-20%. Use of osmotic therapy in such patients has been recommended in both ENLS guidelines for management of intra-cerebral hemorrhage and AHA/ASA guidelines. <sup>13</sup>

Mannitol, is a polyol (sugar and alcohol) a hyper-osmolar agent that has been used for osmotherapy in neurosurgical patients since many years. The proposed mechanism of its action are transient hypervolemia thus decreasing blood viscosity, increase in CBF and the microvascular circulation leading to autoregulatory vasoconstriction and thus reducing cerebral blood volume. However there is controversy regarding its mechanism of effect when given as single bolus dose. Its effect in red blood cell rheology and improved oxygen delivery/circulation has also been hypothesized for explaining its immediate effect in decreasing ICP<sup>14</sup>. Another hypothesis argues about the ability of Mannitol to lower intracranial pressure by reducing brain water content (diuretic effect)<sup>9</sup> and decreasing CSF production.

Pharmacokinetics of Mannitol: Onset of action: 15 minutes Half life: 100 minutes

Osmolarity: 1100 for 20% Mannitol Duration of action: 3-6 hours

Excretion: Urine (80%)

Time of peak action: 30-100 minutes

#### Literature review:

Launey et. al,<sup>15</sup> performed a study to determine the rate of ONSD variation after Mannitol administration for increased ICP episodes. They included thirteen patients in their study comparing and correlating the changes in ONSD, pulsatility index and invasively monitored ICP. The ONSD significantly decreased after Mannitol infusion from 6.3 to 5.56mm (p=0.0007). Concomitantly the intracranial pressure also decreased for 35(32-41) to 25(22-29)mmHg (p=0.001) and the CPP increased from 47 to 69 (p=0.003). The study concluded that the variations of ONSD appear to be an interesting and effective parameter to evaluate the efficacy of osmotherapy for elevated ICP episodes in patients with acute brain injury/SAH.

A study by Li-juan Wang et al<sup>16</sup> which included 60 patients who underwent measurement of ONSD prior to lumbar puncture on admission and during follow up, concluded that ICP was strongly correlated with ONSD(r=0.758, p<0.001) and this association was independent of all other factors like age, sex, BMI, mean arterial pressure and diastolic blood pressure. It also states that ultrasonographic ONSD measurements provide a potential noninvasive method to quantify ICP that can be conducted at the bedside.

Another study performed in the Indian population by Shirodkar et. al<sup>17</sup> evaluated the efficacy of ONSD by ultrasonography as a non-invasive method for detecting raised intracranial pressure in intensive care unit to compare with CT/MRI findings of raised ICP and to prognosticate ONSD value with treatment. The results showed a sensitivity of detecting raised ICP by ONSD to be 84.6% and a specificity approaching around 99%.

A study by Joushua E Nash et al<sup>18</sup> uses ONSD to diagnose raised ICP along with correlation with CT findings. It also reviews the literature from the past and concludes that <0.50 cm ONSD ensured normal pressure (95% CI 0.469-0.540, p<0.001). The study also quantifies the inter-observer variability in ONSD measurement (0.001-0.002cm). The study also determines the expertise required for measuring ONSD to be around 10-25 case examinations and this has been supported by various other studies.

In a prospective convenience sample study, Shushrutha Hedna MD, and colleagues<sup>19</sup> enrolled 86 patients with stroke from a tertiary care center. They measured ONSD on the day of admission and subsequent day, taking longitudinal and transverse measurements of both eyes of each patient. Compared with patients who survived, those who died had increased ONSD in both ischemic stroke categories (0.582 vs. 0.533; P=.0092) and the intracerebral hemorrhage category (0.623 vs. 0.572; P=.0187). With each ONSD increase of 0.1 cm, the odds of mortality increased 4.239 times among patients with ischemic stroke (95% CI, 1.317-13.642; P=.0155) and 6.222 times among patients with intracerebral hemorrhage (95% CI, 1.160-33.382; P=.0329).

Rajajee et al.  $^{20}$  performed a prospective blinded observational study on 65 patients in the ICU. All patients in the study had either had an EVD or intra-parenchymal ICP monitor in situ. The authors used individual as well as mean ONSD values to account for possible fluctuation in the ICP during ONSD measurement. For the individual ONSD measurements the median was 0.53 cm for ICP > 20 mmHg, and was 0.4 cm for ICP < 20 mmHg (p < 0.0001). An ONSD of 0.48 cm demonstrated a sensitivity of 96% and specificity of 94% for predicting ICP > 20 mmHg.

Using a described ONSD cut-off of 5 mm, Tayal et al.<sup>21</sup> performed a prospective blinded observational study in the emergency department on 59 adult patients with a mean age of 38 years, suspected of having raised ICP. The mean ONSD in patients with CT evidence of raised ICP was 6.37 mm, and in the group without evidence of raised ICP, the mean ONSD was 4.94 mm. Using 5 mm as a cut-off point, the study described a sensitivity of 100%, and specificity of 63% for predicting raised ICP.

The use of ONSD measurement specifically in the acute phase (within 6 hours) to detect intracranial haemorrhage (ICH), was investigated by Skoloudik and colleagues<sup>22</sup>. This study included 31 patients with ICH, comparing them to 31 control patients. Sonographic ONSD measurements were performed at 3 and 12 mm behind the globe. Relative ONSD enlargement of > 0.66 mm (> 21%) demonstrated an accuracy of 90.3% for predicting an ICH volume > 2.5cm<sup>3</sup>. The authors then used an ONSD value of > 5mm, demonstrating a sensitivity of 0.708 (95% CI 0.620 – 0.708), specificity of 1.000 (0.697 – 1.000), positive predictive value of 1.000 (95% CI 0.875 – 1.000) and a negative predictive value of 0.500(0.348 – 0.652), concluding that enlargement of the ONSD may be detectable in the hyperacute stage of increased ICP. The use of ONSD to evaluate the clinical evolution of ICH beyond the acute stage was also later confirmed.

A study by Jun IJ and friends<sup>23</sup> aimed at studying the effect of mannitol on ONSD as a surrogate for intracranial pressure during robot assisted laparoscopic prostatectomy with pneumo-peritoneum and the tredelenburg position. Mannitol (0.5 g/kg) was administered after pneumoperitoneum establishment and shifting to the Trendelenburg position. ONSDs were measured at six predetermined time points: 10 minutes after anesthesia induction (T0); 5 minutes after pneumoperitoneum and the Trendelenburg position before Mannitol administration (T1); 30 minutes (T2), 60 minutes (T3), and 90 minutes (T4) after completion of Mannitol administration during pneumoperitoneum and the Trendelenburg position; and at skin closure in the supine position (T5). Results showed that ONSDs were significantly lower at T2, T3, and T4 than at T1 (all p < 0.001), with the greatest decrease observed at T4 compared with T1 (4.46  $\pm$  0.2 mm vs 4.81  $\pm$  0.3 mm, p < 0.001) while mean arterial blood pressure and heart rate were also significantly different. However regional cerebral oxygen saturation, cardiac output, corrected flow time, peak velocity, body temperature, arterial CO<sub>2</sub> partial pressure, peak airway pressure, plateau airway pressure, dynamic compliance, and static compliance were not significantly different during pneumoperitoneum and the Trendelenburg position.

## 4. Rationale and Justification of Study

Optic nerve sheath diameter measurement is a common acute care sonographic procedure. Since the change in intracranial pressure is a continuum of event, sonographic monitoring of such an event is possible through optic nerve sheath diameter monitoring. Mannitol is a common drug used in patients/subjects with raised intracranial pressure either due to trauma, subarachnoid haemorrhage or stroke. Its effects on intracranial pressure reduction are well known though the mechanism is not properly understood yet. My study/research aims at studying the pattern and extent of change in the optic nerve sheath diameter after osmotherapy with intravenous 20% Mannitol within its time of peak effect. Monitoring such changes can help tailor the treatment modality and tier according to efficacy. In absence of invasive monitoring in a limited setup like ours and in light of the various complications associated with invasive monitoring, noninvasive monitoring can help us in improving the outcomes in such neurosurgical or neurological cases.

# 5. Objectives

#### General:

To study the effect of intravenous administration of 20% Mannitol on the optic nerve sheath diameter in patients with raised intracranial pressure.

#### Specific:

- To compare the changes in optic nerve sheath diameter brought about by administration of Mannitol within the time of its peak effect.
- To correlate and compare the extent of change in ONSD ( $\Delta$ ONSD) at 30, 60 and 120 minutes in relation with dose of mannitol administered and change in Mean Arterial Pressure ( $\Delta$ MAP).
- To correlate the changes in ONSD in relation with PIP and PEEP in patients on Mechanical ventilation.

# 6. Research Questions/Hypothesis:

Null Hypothesis ( $H_0$ ): Serial Optic nerve sheath diameter monitoring with a cut-off value of 5.0 mm can reflect changes due to IV administration of 20% Mannitol in patients with raised ICP.

Alternate Hypothesis (H<sub>1</sub>): Serial Optic nerve sheath diameter monitoring with a cut-off value of 5.0 mm cannot reflect changes due to IV administration of 20% Mannitol in patients with raised ICP.

Expected outcome:  $H_0 \neq H_1$ 

# 7. Research Design and Methodology

# 7.1. Research Method

Quantitative

# 7.2 Types of study

Prospective, observational, cross-sectional

# 7.3 Study Population:

All adults in the intensive care unit admitted with the diagnosis of Traumatic brain injury, SAH and acute stroke under treatment with IV 20% Mannitol.

# 7.4 Study site and its justification: Intensive care unit of TUTH, IOM.

Optic nerve sheath diameter has been used for the evaluation of patients with neurological lesion or injuries and in acute care settings. However no studies have been performed on its usefulness in our institute. It can be used to guide the treatment of acute episodes of raised intracranial pressure in the intensive care units and to quantify the efficacy of measures taken to reduce raised intracranial pressure. The examination is easy and is non-interventional, so examination can be made mandatory in such cases.

# 7.5 Sampling Method

Probability sampling

# 7.6 Sample size

Basis and method of determination including power of the study, level of significance etc.

Power of study: 80% (1- $\beta$  = 0.84) Level of significance: 95% ( $\alpha$  = 0.05)

Assuming mean difference and standard deviation of differences ( $\sigma$ ) of 0.24 and 0.49 respectively, effect

size ( $\Delta$ ) was 0.49 as derived from previous study<sup>23</sup>,

Using the formula

$$N = \frac{(z_{1-\alpha/2} + z_{1-\beta})^2}{\Delta^2} + \frac{z_{1-\alpha/2}^2}{2},$$

The sample size required would be 35.

Assuming a dropout of 10%, the required sample size would be 40.

#### 7.7 Inclusion and Exclusion Criteria

# **Inclusion criteria:**

- Age > 18 yrs
- Gender: any
- H/o traumatic brain injury/ subarachnoid hemorrhage/ acute stroke
- Mean optic nerve sheath diameter > 5 mm (0.5 cm)
- Under osmotherapy with 20% Mannitol.

# **Exclusion criteria:**

- Baseline ocular pathology like tumors, Grave's disease and Sarcoidosis
- Previous ocular surgery
- Decompressive cranial surgery

# 7.8 Study Variables:

Epidemiological variables:

Age

Gender

Weight

BMI

# Measured base line variables:

GCS score

Mean arterial pressure

Optic nerve sheath diameter,  $T_1$  (mean of 3 measurements in each eye)

Ventilator parameters (PIP and PEEP) in patients on mechanical ventilation.

# Measured variables after infusion of 20% Mannitol:

Dose of 20% mannitol administered

Mean arterial pressure

Optic nerve sheath diameter (mean of 3 measurements in each eye) after  $30mins(T_2)$ ,  $60 mins(T_3)$  and  $120 mins(T_4)$ .

#### 7.9 Primary outcomes:

Change in the optic nerve sheath diameter ( $\Delta$ ONSD) at  $T_2$ ,  $T_3$  and  $T_4$ .

# 7.10 Secondary outcomes:

Change in the mean arterial pressure before and after mannitol administration.

Comparison and correlation between the extent of change in ONSD ( $\Delta$ ONSD) with dose of mannitol and change in MAP( $\Delta$ MAP).

Correlation between AONSD with PIP and PEEP in mechanically ventilated patients

# 7.10 Expected Duration of the Study: 6 months

# 7.11 Tools and techniques for data collection:

Tools:

6-10 Hz linear array USG probe (Sonosite M-Turbo)

Ultrasound coupling jelly

Transparent dressing (Tegaderm)

Cleaning gauze pieces

Proforma

Arterial blood pressure monitor (invasive or non-invasive)

# Methodology:

- Included patients will be those above 18 years, admitted in the ICU of TUTH, Maharajgunj, with the diagnosis of traumatic brain injury, acute stroke or intracranial hemorrhage and under osmotherapy with 20% Mannitol.
- Written informed consent will be taken from the patient or patient's responsible guardian. Conscious patients will be explained about the procedure.
- The patient's diagnosis, epidemiological variables and baseline variables will be recorded.
- Baseline ventilator parameters will be noted and the ICU staffs instructed not to change those variables over the study period until deemed necessary by the treating physician.
- Positioning of the patient will be done: supine, 30° head elevated.
- Mean arterial blood pressure will be noted from arterial line readings or NIBP reading as appropriate or available.
- A protective transparent dressing will be placed over the closed eyelid in sedated or ventilated patients as an additional measure to prevent any irritation of the conjunctiva.
- For ONSD measurement, generous amount of coupling gel will be applied over the closed upper eyelid.
- The probe will be held with a pincer grasp between the thumb and index finger, using the remaining fingers for stability by resting them on the maxilla or supraorbital ridge.
- The depth will be adjusted to optimize the visualization of the intended structures, i.e. the optic nerve, the surrounding CSF space and the ONS. The gain will be adjusted to create a hypoechoic posterior chamber.
- The mechanical index will be adjusted as per the recommended values for the eye, in order to limit the amount of energy absorbed by the eye.
- Values will be noted 0.3 cm posterior to the retinal surface after optimal visualization of the entry of optic nerve in the orbit.

- Mean will be obtained after taking 3 readings in each eye. Only patients with mean ONSD > 0.5cm will be included and the baseline value designated as T<sub>1</sub>.
- Intravenous 20% Mannitol as prescribed will be administered via a dedicated IV line over 20 minutes.
- Mean arterial pressure and Optic nerve sheath diameter readings will be performed as previously described and noted at  $30(T_2)$ ,  $60(T_3)$  and  $120(T_4)$  minutes after completion of IV administration.
- The coupling gel will be removed gently after each measurement and the protective adhesive dressing will be removed at the end of the study.

# 7.12 Management protocol of patients/participants if applicable:

All patients will be managed according to the current ICU protocol abiding with the ENLS and Brain Trauma Foundation guidelines for TBI and intra-cerebral hemorrhage and AHA/ASA guidelines for acute ischemic stroke. In subjects with persistently elevated intracranial pressure and ONSD findings above 5.0 mm despite the administration of 20% Mannitol, decision for further treatment will rest upon the treating physician.

# 7.13 Plan for Data Management and Statistical Analysis

- Data will be entered by the investigator and resident on duty in the intensive care unit and will be destroyed after the completion of the study, however the results and conclusions will be stored without hampering the subject/ patient's privacy or rights.
- Power of the study is based on the primary outcome which is the change in ONSD following infusion of 20% Mannitol.
- Paired t test, chi square test will be used for data analysis.
- Data will be analysed by using SPSS 20 software version
- The value of p<0.05 will be considered as statistically significant.

# 7.14 A graphic outline of the study design and procedures using a flow diagram including the timing of assessments.



# 8. Biases:

Data collection by on duty MD anesthesiology Resident or DM Critical Care Residents will reduce observer and performance bias.

# 9. Limitation of the study:

Single centered Open label No control group

# 10. Safety considerations:

Regarding the safety concerns during the measurement of optic nerve sheath diameter subjects with ocular injury, glaucoma are being excluded. The acoustic energy used for diagnostic purposes has no described adverse effects. The recent bioeffects and safety report by the American Institute of Ultrasound in Medicine (AIUM) makes no specific mention of the eye. The United States Food and Drug Administration Center for Devices and Radiological Health (US FDA/CDRH) describes an output intensity limit for all eye exposure of 50 mW/cm2, recommending the use of a mechanical index (MI) < 0.23, and a thermal index (TI) < 1. The definition of an experienced operator differs, but studies have defined an experienced operator as having performed more than 25 prior transorbital ultrasound examinations.

# 11. Plan for Supervision and Monitoring:

The research will be continuously supervised by the co-guides Dr. Pramesh Sundar Shrestha and Dr. Arjun Gurung and will be conducted under the guidance of Dr. Subhash P. Acharya.

# 12. Expected outcome of the Research:

Optic nerve sheath diameter changes are expected to be associated with the administration of 20% Mannitol in patients with raised intracranial pressure. Such an outcome would have various benefits in terms of usefulness of the optic nerve sheath diameter monitoring.

#### 13. Plan for Dissemination of Research:

Research results will be submitted to the Department of Anaesthesiology and Research department, IOM.

Research results will also be submitted for publication in national and international journals of repute.

#### 14. Plan for Utilization of the Research Findings:

The research results would help us in the care of patients in the neurosurgical and neurological intensive care units with non-invasive monitoring.

# 15. Work Plan

| S.N | Activities | 2018 AD | | 2019 AD | | | |
|---|---|---|---|---|---|---|---|
| | | Nov | Dec | Jan | Feb | Mar | Apr |
| 1 | Problem identification | | | | | | |
| 2 | Literature review | | | | | | |
| 3 | Topic selection | | | | | | |
| 4 | Writing thesis proposal | | | | | | |
| 5 | Presentation to sub committee | | | | | | |
| 6 | Review thesis proposal | | | | | | |
| 7 | Submission to IRB | | | | | | |
| 8 | Approval from IRB | | | | | | |
| 9 | Data collection | | | | | | |
| 10 | Data analysis | | | | | | |
| 11 | Final thesis writing | | | | | | |
| 12 | Final correction and submission | | | | | | |

# 16. Ethical Consideration

Research is based on human optic nerve sheath diameter.

Approval by IRB.

Verbal consent from patients relatives and/or legal guardian would suffice as the study is non-interventional and non-invasive with no effect on patients safety.

Confidentiality will be maintained.

# 17. Obtaining the Consent

Patients legal guardian will be well counseled and no information will be withheld.

# 18. Budget

The expenditure during the study will be made by the principal investigator.

Transparent dressing (Tegaderm): 50 pcs: Rs. 2400

Data statistician: Rs. 8000 Stationary: Rs. 4000

Photocopies of proforma and information sheet: Rs.2000

Binding: Rs. 4000 Total: Rs 20400

#### 19. Annexes:

Date:\_\_\_\_/\_\_\_\_

#### INFORMED CONSENT

Department of Anaesthesiology

Tribhuvan University, Institute of Medicine, Kathmandu, Nepal,

Study Title: Effect of intravenous administration of Mannitol 20% on the Optic nerve sheath diameter(ONSD) in patients with raised intracranial pressure Subject's Initials: Study Number: Subject's Name: Date of Birth / Age: \_\_\_\_\_ (i) I confirm that I have read and understood the information sheet and consent form dated for the above study and have had the opportunity to ask questions. (ii) I understand that my participation in the study is voluntary and that I am free to withdraw at any time, without giving any reason, without my medical care or legal rights being affected. (iii) I understand that the researchers and the IRB and other regulatory authorities will not need my permission to look at my health records both in respect of the current study and any further research that may be conducted in relation to it, even if I withdraw from the trial. I agree to this access. However, I understand that my identity will not be revealed in any information released to third parties or published. (iv)I agree not to restrict the use of any data or results that arise from this study provided such a use is only for scientific purpose(s) (v) I agree to take part in the above study. Signature (or Thumb impression) of the Subject/Legal Guardian: Signature of the Investigator: Signatory's Name: Date:\_\_\_\_/\_\_\_\_ Study Investigator's Name: Date:\_\_\_/\_\_\_/ Signature of the Witness: Name of the Witness:

# सुसूचित मन्जुरीनामा

| म | | (उमेर | वर्ष)ले | Study on | the effec | et of |
|---|---|---|---|---|---|---|
| intravenous adminis | | | | | | with |
| raised intracranial ] | pressure' शिर्षक | को अनुसन्धान स | म्बन्धी संलग्न | मिति २०७ | / / | को |
| 'जानकारी पत्र/पुसि | -तका' सुनेर/पढे | र र प्रश्नोत्तर समेत | गरेर यो अध्यय | ग्न-अनुसन्ध | ान सम्बन | धमा |
| जानकारी प्राप्त भ | यो। यो अनुसन्ध | ान कार्यमा मेरो स | हभागिता मेरो व | यक्तिगत इ | च्छामा भ | र पर्ने |
| र मैले चाहेको खण | डमा कुनै पनि बे | ला यो अनुसन्धान | प्रक्रियाबाट बार्गि | हेरिन पाउने | भन्ने कुरा | मैले |
| बुझेको छु। यसको | लागि मैले कुनै | कारण दिनु नपर्ने | र त्यसबाट मैले | पाउने सेवा | र मेरो क | ानुनी |
| अधिकारमा असर | नपर्ने समेत मल | ाई बुझाईएकोछ। र | यस अनुसन्धान | को प्रतिवेदन | वा सम्बर्गि | न्धत |
| प्रकाशित कृतिहरु | ना मेरो कुनै र्व्या | क्तगत परिचय खु | ल्ने जानकारी प्र | काशित हुने | छैन भन्ने | कुरा |
| मैले बुझेकोछु। | | | | | | |
| सहभागीको बुढीओ | लाको ल्याप्चे | | | | | |
| U | <b></b> | | | | | |
| दायाँ | बायाँ | | | | | |
| यी सबै कुराहरु जा | नी-बुझी, म यस | अध्ययन-अनुसन | धानमा सहभागी | हुन स्वेच्छा | ले राजी भ | ई यो |
| सुसूचित मन्जुरीन | ामामा सहिछाप | गरेकोछु। | | | | |
| सहभागीको सही_ | | | | | | |
| सहभागीको नाम १ | गर | | | | | |
| मिति २०७ / / | | | | | | |
| साक्षीको सही | | | | | | |
| साक्षीको नाम थर | | | | | | |

# **Proforma**

"Study on the effect of intravenous administration of 20% Mannitol on the Optic nerve sheath diameter (ONSD) in patients with episodes of raised intracranial pressure."

| Participant serial no.: | IP no.: | Date: |
|-------------------------|-----------------|---------|
| Name: | Age/sex: | Weight: |
| Height: | BMI: | |
| Diagnosis: | Admission date: | |

Ventilator parameters at time of baseline measurement

PIP:  $cmH_2O$ 

PEEP: cmH<sub>2</sub>O

Time of 20% Mannitol administration: Dose of 20% Mannitol administered: Time of measurement: 30 minutes:

60 minutes: 120 minutes:

#### MEASURED VARIABLES:

| MEASURED VARIABLES. | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| VARIABLES BASELINE | | POST-MANNITOL | | 60 MINUTE | | 120 MINUTES | | | |
| | | $(T_1)$ | | (30MINUT | <b>ES: T2)</b> | $(T_3)$ | | $(T_4)$ | |
| MEAN | | | mmHg | | mmHg | | mmHg | | mmHg |
| ARTERIAL | , | | | | | | | | |
| PRESSURE | ·<br>/ | | | | | | | | |
| OPTIC 1 | NERVE | RIGHT: | mm | RIGHT: | mm | RIGHT: | mm | RIGHT: | mm |
| SHEATH | | LEFT: | mm | LEFT: | mm | LEFT: | mm | LEFT: | mm |
| DIAMETER | } | MEAN: | mm | MEAN: | mm | MEAN: | mm | MEAN: | mm |
| GLASGOW | 7 | E: | | E: | | E: | | E: | |
| COMA SCA | <b>ALE</b> | V: | | V: | | V: | | V: | |
| | | M: | | M: | | M: | | M: | |

# **List of Abbreviations:**

| ICP | Intracranial pressure |
|---|---|
| TBI | Traumatic brain injury |
| SAH | Subarachnoid hemorrhage |
| ONSD | Optic nerve sheath diameter |
| СРР | Cerebral perfusion pressure |
| CBF | Cerebral Blood Flow |
| MAP | Mean arterial pressure |
| GCS | Glasgow Coma Scale |
| USG | Ultrasonography |
| ICU | Intensive care unit |
| IOM | Institute of medicine |
| TUTH | Tribhuwan University Teaching Hospital |
| IV | Intravenous |
| BMI | Body Mass Index |
| ASA/AHA | American Heart Association/American Stroke<br>Association |
| SPSS | Statistical Package for the Social Sciences |
| TCD | Transcranial Doppler |
| cmH <sub>2</sub> O | Centimeter of water |
| COR | Class of recommendation |
| LOE | Level of evidence |
| MI | Mechanical index |
| TI | Thermal index |
| US FDA/CDRH | United States Food and Drug Administration/<br>Center for Devices and Radiological Health |
| AIUM | American Institute Of Ultrasound In Medicine |
| ENLS | <b>Emergency Neurological Life Support</b> |
| CI | Confidence Interval |
| PIP | Peak Inspiratory Pressure |

#### REFERENCES:

- 1. Miller JD, Sullivan HG. Severe intracranial hypertension. Int Anesthesiol Clin. 1979;17(2-3):19-75.
- 2. Rangel-Castilla, L., Gopinath, S. & Robertson, C. S.. 2008. Management of intracranial hypertension. Neurol Clin 26: 521-41, x. doi: 10.1016/j.ncl.2008.02.003.
- 3. Geeraerts T, Launey Y, Martin L, Pottecher J, Vigué B, Duranteau J, et al. Ultrasonography of the optic nerve sheath may be useful for detecting raised intracranial pressure after severe brain injury. Intensive Care Medicine. 2007Jan;33(10):1704–11
- 4. Legrand A, Jeanjean P, Delanghe F, Peltier J, Lecat B, Dupont H. Estimation of optic nerve sheath diameter on an initial brain computed tomography scan can contribute prognostic information in traumatic brain injury patients. Critical Care. 2013;17(2)
- 5. Chesnut RM, Temkin N, Carney N, et al. A Trial of Intracranial-Pressure Monitoring in Traumatic Brain Injury. The New England journal of medicine. 2012;367(26):2471-2481. doi:10.1056/NEJMoa1207363.
- 6. Williams P. Optic Nerve Sheath Diameter as a Bedside Assessment for Elevated Intracranial Pressure. Case Reports in Critical Care. 2017;2017:1–2
- 7. Kimberly H, Shah S, Marill K, Noble V. Correlation of Optic Nerve Sheath Diameter with Direct Measurement of Intracranial Pressure. Academic Emergency Medicine. 2007Jan;14 (5 Supplement 1).
- 8. Soldatos T, Karakitsos D, Chatzimichail K, Papathanasiou M, Gouliamos A, Karabinis A. Optic nerve sonography in the diagnostic evaluation of adult brain injury. Crit Care. 2008;12(3):R67.
- 9. Diringer MN, Scalfani MT, Zazulia AR, Videen TO, Dhar R, Powers WJ. Effect of mannitol on cerebral blood volume in patients with head injury. Neurosurgery. 2012;70(5):1215-8; discussion 9.
- 10. Hlatky R, Valadka AB, Robertson CS. Intracranial hypertension and cerebral ischemia after severe traumatic brain injury. Neurosurg Focus. 2003;14(4):e2.
- 11. Carney N, Totten AM, O'Reilly C, Ullman JS, Hawryluk GW, Bell MJ, et al. Guidelines for the Management of Severe Traumatic Brain Injury, Fourth Edition. Neurosurgery. 2017;80(1):6-15.
- 12. Zoerle T, Lombardo A, Colombo A, Longhi L, Zanier ER, Rampini P, et al. Intracranial pressure after subarachnoid hemorrhage. Crit Care Med. 2015;43(1):168-76.

- 13. Powers WJ, Rabinstein AA, Ackerson T, Adeoye OM, Bambakidis NC, Becker K, et al. 2018 Guidelines for the Early Management of Patients With Acute Ischemic Stroke: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2018;49(3):e46-e110.
- 14. Sakowitz OW, Stover JF, Sarrafzadeh AS, Unterberg AW, Kiening KL. Effects of mannitol bolus administration on intracranial pressure, cerebral extracellular metabolites, and tissue oxygenation in severely head-injured patients. J Trauma. 2007;62(2):292-8.
- 15. Launey Y, Nesseler N, Le Maguet P, Malledant Y, Seguin P. Effect of osmotherapy on optic nerve sheath diameter in patients with increased intracranial pressure. J Neurotrauma. 2014;31(10):984-8.
- 16. Wang LJ, Chen LM, Chen Y, Bao LY, Zheng NN, Wang YZ, et al. Ultrasonography Assessments of Optic Nerve Sheath Diameter as a Noninvasive and Dynamic Method of Detecting Changes in Intracranial Pressure. JAMA Ophthalmol. 2018;136(3):250-6. doi: 10.1001/jamaophthalmol.2017.6560.
- 17. Shirodkar CG, Rao SM, Mutkule DP, Harde YR, Venkategowda PM, Mahesh MU. Optic nerve sheath diameter as a marker for evaluation and prognostication of intracranial pressure in Indian patients: An observational study. Indian J Crit Care Med. 2014;18(11):728-34.
- 18. Nash, J. E., O'Rourke, C., & Moorman, M. L. (2016). Transocular ultrasound measurement of the optinerve sheath diameter can identify elevated intracranial pressure in trauma patients. *Trauma*, *18*(1),28–34. https://doi.org/10.1177/1460408615606752
- 19. Shushrutha Hedna, Vishnumurthy, Rastogi, Vaibhav, Weeks, Emily & Patel, Rohit P. 2015. Abstract WMP83: Use of Optic Nerve Sheath Diameter in Emergency Department to Predict Stroke Outcome. Stroke 46: AWMP83-AWMP83.
- 20. Rajajee V, Vanaman M, Fletcher JJ, Jacobs TL. Optic nerve ultrasound for the detection of raised intracranial pressure. Neurocrit Care. 2011;15(3):506-15.
- 21. Tayal VS, Neulander M, Norton HJ, Foster T, Saunders T, Blaivas M. Emergency department sonographic measurement of optic nerve sheath diameter to detect findings of increased intracranial pressure in adult head injury patients. Ann Emerg Med. 2007;49(4):508-14.
- 22. Skoloudik D, Herzig R, Fadrna T, Bar M, Hradilek P, Roubec M, et al. Distal enlargement of the optic nerve sheath in the hyperacute stage of intracerebral haemorrhage. Br J Ophthalmol. 2011;95(2):217-21.
- 23. Jun I-J, Kim M, Lee J, Park S-U, Hwang J-H, Hong JH, et al. Effect of Mannitol on Ultrasonographically Measured Optic Nerve Sheath Diameter as a Surrogate for Intracranial Pressure During Robot-Assisted Laparoscopic Prostatectomy with Pneumoperitoneum and the Trendelenburg Position. J Endourol. 2018 Jul;32(7):608–13.